CLINICAL TRIAL: NCT06297538
Title: Targeting the Motor Cortex in Parkinson's Disease by Gamma-transcranial Alternating Current Stimulation: Pathophysiological and Therapeutic Implications
Brief Title: Parkinson's Disease and Gamma-transcranial Alternating Current Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromed IRCCS (Other)
Collaborators: Fondazione Policlinico Universitario Campus Bio-Medico (Other); I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Giulia Paparella, Principal Investigator, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR-2021-12372323
Record Dates: First submitted 2024-02-22; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Motor cortex; Transcranial magnetic stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gamma transcranial alternating current stimulation (Experimental)
  Interventions: Device: gamma transcranial alternating current stimulation (tACS)
- sham transcranial alternating current stimulation (Sham Comparator)
  Interventions: Device: sham transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Device: gamma transcranial alternating current stimulation (tACS) — Transcranial alternating current stimulation (tACS) will be delivered using a BrainSTIM (EMS, Italy) connected to two electrodes (5x5cm) enclosed in sponges soaked with saline solution. One electrode will be centred over the first dorsal interosseus (FDI) hotspot and the other over P3. tACS will be delivered at peak-to-peak amplitude of 1 milliampere (mA), and with 3-seconds ramp-up and down periods. The stimulation frequency will be 70 Hz, as representative of the endogenous motor network-related gamma frequency.
  Arms: gamma transcranial alternating current stimulation
Device: sham transcranial alternating current stimulation (tACS) — Sham-tACS will consist of ramp-up and down periods and only 1-second stimulation at 1 mA amplitude.
  Arms: sham transcranial alternating current stimulation

SUMMARY:
Cortical-basal ganglia gamma oscillations are pathologically reduced in Parkinson's disease (PD) and the plasticity of the primary motor cortex (M1) is impaired. Enhancing gamma oscillations through transcranial alternating current stimulation (tACS), a non-invasive neurophysiological tool that modulates cortical rhythms, can restore this alteration. However, whether tACS-related normalization of M1 plasticity results in positive clinical effects is unknown. Motor learning is also impaired in PD and gamma oscillations play a relevant role in different forms of learning in humans. Nevertheless, whether motor learning abnormalities relate to reduced gamma oscillations in PD is another unclear issue. It can be hypothesized that gamma oscillations impairment in M1 contributes to altered motor control, plasticity and learning in PD. Accordingly, in this project, the authors intend to test whether gamma-tACS on M1 in PD patients ameliorates motor performance and learning, as objectively assessed with kinematic techniques.

ELIGIBILITY:
Inclusion Criteria:

* PD diagnosis

Exclusion Criteria:

* severe cognitive and psychiatric comorbidities
* H&Y>3
* levodopa-induced dyskinesia and tremor-dominant phenotype
* history of additional neuropsychiatric disorders
* intake of medications acting on brain excitability or plasticity
* contraindications to non-invasive brain stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-04-29 (Actual); Primary Completion 2024-10-29 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Changes in bradykinesia features as objectively assessed by kinematic techniques | post 5, 15 and 30 minutes
  The velocity of finger tapping movements will be kinematically measured and expressed in degrees/second.
Changes in motor learning performance as objectively assessed by kinematic techniques | post 5, 15 and 30 minutes
  The acceleration peak of finger index abductions will me kinematically measured and expressed as millimeters/seconds

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, Italy

IPD SHARING:
Plan to Share IPD: No